CLINICAL TRIAL: NCT03927846
Title: Web-based Pain Self-Management: Nurse-Guided
Brief Title: Implementation of Nurse-guided Web-based Cognitive Behavioral Therapy for Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00056912; UL1TR001420 (NIH)
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Results first posted 2021-07-15 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2021-02

CONDITIONS: Chronic Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Participants (n=60) in the primary care and rheumatology clinics will be randomized to one of 2 arms: (1) 6 regular telephone contacts, vs. (2) 6 computer generated email reminders (control arm) over an 8-week period. To enhance participants' motivation to engage in the web-based CBT, nurses will use motivational interviewing technique.
Who Masked: Outcomes Assessor
Masking Description: Study coordinator will be blinded to randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone Contact (Nurse) (Active Comparator): 6 regular telephone contacts by nurses who will use a motivational interviewing technique
  Interventions: Behavioral: Nurse-guided Web-based Cognitive Behavioral Therapy
- E-mail contact (Active Comparator): 6 computer generated email reminders (control arm) over an 8-week period.
  Interventions: Behavioral: Nurse-guided Web-based Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Nurse-guided Web-based Cognitive Behavioral Therapy — nurse contact is to support and enhance participants' motivation to engage in the web-based CBT program.

SUMMARY:
To see if nurse guided web based cognitive behavioral therapy (CBT) will show pain improvement in patients with all types of pain complaints.

DETAILED DESCRIPTION:
The primary objective of this application is to test the feasibility of a care model where clinic nurses play a vital role in promoting the adoption of web-based CBT in the ambulatory medical setting. Participants (n=60) in the primary care and rheumatology clinics will be randomized to one of 2 arms: (1) 6 regular telephone contacts, vs. (2) 6 computer generated email reminders (control arm) over an 8-week period. To enhance participants' motivation to engage in the web-based CBT, nurses will use motivational interviewing technique. The investigators will use outcome measures including the number of completed web-based learning modules, amount of time spent by the nurses on study-related and non-study related phone calls, health care use, and clinical variables. Our proposed line of research is significant because it will potentially make CBT, a significantly underutilized treatment modality, potentially more affordable and accessible. If nurse guided web-based CBT can be shown to be effective and implementable, Wake Baptist Health System can potentially leverage web-based CBT as one component in a multidisciplinary pain management program to prospective employers in North Carolina. Wake Baptist may also develop its own web-based CBT for commercial use.

ELIGIBILITY:
Inclusion Criteria: -

1. patients at the primary care or rheumatology clinic with daily pain for 6 months or longer affecting the low back, neck, hip, knee or widespread pain;
2. at least moderate in average pain severity, defined as a weekly average pain severity score of 5 or greater 24;
3. at least 18 years of age;
4. reliable phone (landline or cell), and
5. have home computer with reliable internet access.

Exclusion Criteria:

1. planned elective surgery during the study period;
2. very severe symptoms of depression (i.e., The eight-item Patient Health Questionnaire depression scale (PHQ8) score of ≥ 20);
3. ongoing unresolved disability claims;
4. inflammatory arthritis (e.g., lupus, rheumatoid arthritis, ankylosing spondylitis, etc.);
5. cancer-related musculoskeletal pain;
6. history of bipolar disorder or schizophrenia; and
7. takes daily opioid for more than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Ang, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
If nurse guided web-based CBT can be shown to be effective and implementable, Wake Baptist can potentially leverage web-based CBT as one component in a multidisciplinary pain management program to prospective employers in North Carolina. With assistance from Wake Forest Innovation, Wake Baptist may also develop its own web-based CBT that can be commercialize in the future.

RESULTS

PARTICIPANT FLOW:
Groups:
- Nurse Support: Participants received phone-based coaching
- Control: No contact with the research team
Period: Overall Study
Arm/Group | Nurse Support | Control
Started | 30 | 30
Completed | 20 | 19
Not Completed | 10 | 11
Not completed — Lost to Follow-up | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nurse Support | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (14.9) | 51.8 (20.5) | 52.1 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 49
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 29 | 29 | 58
  Unknown or Not Reported | 0 | 0 | 0
PROMIS pain intensity [Mean (Standard Deviation); unit: units on a scale] — Questionnaire that measures subject pain intensity. The possible score range is 3-15, 3 being the best outcome and 15 being the worst outcome
  units on a scale | 5.8 (1.6) | 6.0 (1.9) | 5.9 (1.7)
PROMIS pain interference [Mean (Standard Deviation); unit: T-Score] — PROMIS pain interference is a questionnaire that measures interference of pain on subject's life. The possible raw score range is 6-30. The raw score has been converted into a T score. The T score range is from 41.6 to 75.6. A t-score indicates the number of standard deviations away from the mean. A t-score of 50 is equal to the mean of a reference population. Values below 50 indicate pain interference better than the reference population and values above 50 indicate pain interference worse than the reference population.
  T-Score | 61.2 (7.4) | 62.9 (6.5) | 62.1 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: PROMIS (Patient Reported-outcomes Measurement Information System) Pain Intensity
Description: Questionnaire that measures subject pain intensity. The possible score range is 3-15, 3 being the best outcome and 15 being the worst outcome
Time Frame: Up to Week 16
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Nurse Support | Control
Number analyzed (Participants) | 20 | 19
score on a scale | 4.4 (0.3) | 4.7 (0.2)

2. Primary Outcome: PROMIS Pain Interference
Description: PROMIS pain interference is a questionnaire that measures interference of pain on subject's life. The possible raw score range is 6-30. The raw score has been converted into a T score. The T score range is from 41.6 to 75.6. A t-score indicates the number of standard deviations away from the mean. A t-score of 50 is equal to the mean of a reference population. Values below 50 indicate pain interference better than the reference population and values above 50 indicate pain interference worse than the reference population.
Time Frame: Up to Week 16
Measure: Mean (Standard Error); unit: T-score
Arm/Group | Nurse Support | Control
Number analyzed (Participants) | 20 | 19
T-score | 57.4 (0.9) | 57.3 (0.9)

3. Secondary Outcome: Completed Phone Calls
Description: The number of completed phone calls by the nurse will be recorded.
Time Frame: Up to Week 16
Measure: Median (Inter-Quartile Range); unit: number of phone calls
Arm/Group | Nurse Support | Control
Number analyzed (Participants) | 20 | 19
number of phone calls | 3.5 [2 to 5] | 0 [0 to 0]

4. Secondary Outcome: Completed Learning Modules Per Treatment Arm
Description: The number of completed learning modules per treatment arm will be recorded.
Time Frame: Week 16
Measure: Median (Inter-Quartile Range); unit: number of learning modules
Arm/Group | Nurse Support | Control
Number analyzed (Participants) | 30 | 30
number of learning modules | 7 [1 to 8] | 8 [1 to 8]

5. Other Pre Specified Outcome: Proportion of Subjects With Interest in Pain Self-management
Description: This refers to the acceptability a subject has to pain self management. This would be determined by the number of subjects who answer "yes" to the question "Have you ever wondered if there is something that you could do on your own to better manage your pain?" divided by the number of patients who answered "yes" to the question "Over the last 6 months, do you have daily or almost daily pain that interfered with your general activity or enjoyment of life?"
Time Frame: Up to Week 16
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Proportion of Patients Who Viewed Educational Video
Description: This refers to the acceptability a subject has to watching the educational video on web-based CBT. This would be determined by the number of patients who watched the video from Expectation Management and Medical Information (EMMI) divided by the number of patients who received the video from EMMI.
Time Frame: Up to Week 16
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Proportion of Subjects Who Called the Research Coordinator to Participate in the Study.
Description: This refers to the acceptability a subject has to participating in the study. This would be determined by the number of patients who made a phone call to the research team after watching the video divided by the number of patients who watched the video.
Time Frame: Up to Week 16
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Ratings of Perceived Disruption
Description: This refers to whether health care personnel perceives a disruption in the clinic standard operating procedures
Time Frame: Up to Week 16
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Uptake Rates
Description: This refers to the adoption or extent of participants' motivation to engage in the web-based CBT program. For the uptake rate, the number of times participants log in to web-based CBT will be recorded.
Time Frame: Up to Week 16
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Self-report Frequency of Practicing Pain Coping Skills
Description: This refers to the adoption or extent of participants' motivation to engage in the web-based CBT program. Self-report frequency of practicing pain coping skills will be measured by a question scale 0-5. Higher scores denote better outcomes.
Time Frame: Up to Week 16
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Participant Overall Satisfaction on Web-based CBT Program
Description: This refers to the adoption or extent of participants' motivation to engage in the web-based CBT program. Recorded in a question - scale 0-5. Higher scores denote better outcomes.
Time Frame: Up to Week 16
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Nurse's Time
Description: This refers to the feasibility of the web-based CBT program. The number of minutes a nurse spends on study-related phone calls and the time a nurse spends during the initial and ongoing MI training will be recorded.
Time Frame: Up to Week 16
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Perceived Work Rating
Description: This refers to the feasibility of the web-based CBT program. Nurses will rate perceived additional work load. Recorded using sing a scale 1-5, higher scores denotes worse outcomes.
Time Frame: Up to Week 16
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Motivational Interviewing Treatment Integrity (MITI) Scale
Description: This refers to the feasibility of the web-based CBT program. This scale is used to assess treatment fidelity to the principles of MI.Scale range from 5 to 25, where a score of 25 represents 100% adherence to the principles of motivational interviewing (MI).
Time Frame: Up to Week 16
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Mean Opioid Daily Dose
Description: This refers to the burden or utilization of health care in relation to the web-based CBT program. The mean daily dose of opioids will be recorded for all participants.
Time Frame: Up to Week 16
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Non-study Phone Calls
Description: This refers to the burden or utilization of health care in relation to the web-based CBT program. The number of pain relevant phone calls will be recorded.
Time Frame: Up to Week 16
Reporting Status: Not Posted

17. Other Pre Specified Outcome: New Referrals to Other Musculoskeletal-related Specialties
Description: This refers to the burden or utilization of health care in relation to the web-based CBT program. The number of new referrals to other musculoskeletal-related specialties will be recorded.
Time Frame: Up to Week 16
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Number of Emergency Room Visits Related to Pain
Description: This refers to the burden or utilization of health care in relation to the web-based CBT program. The number of ER visits per subject related to pain will be recorded.
Time Frame: Up to Week 16
Reporting Status: Not Posted

19. Other Pre Specified Outcome: PROMIS Physical Health -Fatigue
Description: This is a questionnaire that pertains to subject physical health. Raw summed score from 4 to 20, where 20 represents severe fatigue.
Time Frame: Up to Week 16
Reporting Status: Not Posted

20. Other Pre Specified Outcome: PROMIS Physical Health - Physical Function
Description: This is a questionnaire that pertains to subject physical health. Raw summed score from 4 to 20, where 20 represents severe physical impairment.
Time Frame: Up to Week 16
Reporting Status: Not Posted

21. Other Pre Specified Outcome: PROMIS Physical Health - Sleep-related Impairment
Description: This is a questionnaire that pertains to subject physical health.Raw summed score from 4 to 20, where 20 represents severe sleep impairment.
Time Frame: Up to Week 16
Reporting Status: Not Posted

22. Other Pre Specified Outcome: PROMIS Physical Health- Pain Behavior
Description: This is a questionnaire that pertains to subject physical health. Raw summed score from 20 to 100, where 100 represents severely maladaptive pain behavior.
Time Frame: Up to Week 16
Reporting Status: Not Posted

23. Other Pre Specified Outcome: PROMIS Social Health
Description: This is a questionnaire that pertains to subject social health. Raw summed score range from 4 to 20, where 20 represents complete inability to participate in various social functions.
Time Frame: Up to Week 16
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Brief Pain Inventory (BPI) Pain Severity
Description: This is a pain severity questionnaire. BPI consists of four items that are scored from 0 (no pain) to 10 (worst possible pain); the mean of this four areas is reported as the score.
Time Frame: Up to Week 16
Reporting Status: Not Posted

25. Other Pre Specified Outcome: BPI Pain Interference
Description: This is a questionnaire that shows a subject's perceived interference of pain in his/her daily life. The BPI pain interference section consists of seven items that are scored from 0 (no interference) to 10 (complete interference).A pain interference score is calculated from the mean of the seven pain interference items.
Time Frame: Up to Week 16
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Nurse Support | Control
Number analyzed (Participants) | 20 | 19
score on a scale | 3.5 (0.3) | 3.5 (0.3)

26. Other Pre Specified Outcome: Pain Catastrophizing Score (PCS)
Description: This questionnaire shows the subject's perceived pain. The score is from 0-52 with 0 being the best outcome and 52 being the worst outcome.
Time Frame: Up to Week 16
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Global Rating of Change (GRoC)
Description: This questionnaire shows how the subject rates his/her overall condition of pain from the beginning of treatment to when the questionnaire is completed. The score ranges from -5 to 5, with -5 being the worst outcome and 5 being the best outcome.
Time Frame: Up to Week 16
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Patient Health Questionnaire Depression Scale (PHQ-8)
Description: A questionnaire that shows patient's level of depression. Scores can be 0-24, with 0 being the best outcome and 24 being the worst. A score of 10 or greater is considered major depression. A score of 20 or more is severe major depression.
Time Frame: Up to Week 16
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Generalized Anxiety Disorder (GAD-7)
Description: A questionnaire that shows how much anxiety a subject has. Scores can be 0-18. A score of 5-9 means mild anxiety. A score of 10-14 means moderate anxiety. A score of 15-18 means severe anxiety.
Time Frame: Up to Week 16
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Nurse Support | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT03927846/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/46/NCT03927846/SAP_001.pdf
  • Informed Consent Form (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT03927846/ICF_002.pdf